CLINICAL TRIAL: NCT04976127
Title: Safety Evaluation of Intravenous Talineuren (TLN) in Parkinson's Disease-affected Patients
Acronym: NEON
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InnoMedica Schweiz AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TLN/PD/1
Record Dates: First submitted 2021-05-16; First posted 2021-07-26 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Part 1: dose escalation phase, 3 patients with Parkinson's disease, (2 cohorts as in 1+2 patients, sequential inclusion between the first and 2nd patient)
  Part 2: repeated dose administration phase, 9 patients with Parkinson's disease (1 cohort)
  Part 3: Dose consolidation with intrapatient dosing, 10 patients with Parkinson's disease (1 cohort)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Talineuren dose escalation (Experimental): 14 doses of GM1 Ganglioside 6, 12, 60, 120, 180, 240, 300, 360, 420, 480, 540, 600, 660, 720 mg. Optional treatment prolongations for 16 weeks (Amendment 2), 8 months (Amendment 3), 4 months (Amendment 4) and 12 months (Amendment 5).
  Interventions: Drug: Talineuren
- Talineuren repeated dose (Experimental): 8 repeated doses of GM1 Ganglioside tbd from the escalation dose (maximum suitable dose). Optional treatment prolongations for 16 weeks (Amendment 2), 8 months (Amendment 3), 4 months (Amendment 4) and 12 months (Amendment 5).
  Interventions: Drug: Talineuren
- Talineuren dose consolidation with intrapatient dosing (Experimental): 8 months repeated doses of 720mg GM1 Ganglioside (Amendment 3).
  Interventions: Drug: Talineuren

INTERVENTIONS:
Drug: Talineuren — Talineuren is a liposomal formulation of the GM1 Ganglioside for intravenous administration
  Other Names: liposomal GM1

SUMMARY:
This study is an open-label, single ascending dose escalation followed by a multiple administration dose at the maximal suitable dose (MSD). The investigational Medicinal Product (IMP) is given as an add-on therapy.

Talineuren consists of GM1 (monosialotetrahexosylganglioside), the pharmacologically active ingredient, associated with a proprietary lipid formulation assembled as liposomes.

The primary objective is to demonstrate the safety of TLN administration intravenously in Parkinson patients.

Secondary objectives are the determination of the maximal suitable dose based on the safety profile and preliminary efficacy, as well as the determination of the pharmacokinetics (PK) profile.

DETAILED DESCRIPTION:
The ganglioside lipid GM1 has been described in the literature as a neuroprotective agent.

Several clinical studies have shown that GM1 improves the condition of Parkinson's disease patients.

Talineuren consists of the pharmacologically active ingredient GM1, associated with a proprietary lipid formulation assembled as liposomes. Talineuren has been developed to improve the delivery and bioavailability of GM1.

The primary objective of this trial is to demonstrate the feasibility and safety of intravenous Talineuren administration in Parkinson's disease patients.

The secondary objectives are:

* The determination of the recommended phase 2 dose based on the safety profile and preliminary efficacy.
* The determination of the pharmacokinetics (PK) profile.

This trial aims to investigate the safety of the novel formulation of GM1, Talineuren.

To that extent a three-part trial was designed: Part 1- Dose escalation Part 2- Dose consolidation Part 3- Dose consolidation with intrapatient dosing

Part 1- rapid dose escalation scheme from 6 mg to 720 mg of Talineuren formulated GM1 in 3 patients. Optional treatment prolongations for 8 weeks (Amendment 1), 16 weeks (Amendment 2), 8 months (Amendment 3), 4 months (Amendment 4), and 12 months (Amendment 5).

Part 2- multiple dosing of Talineuren over 8 weeks in 9 patients to validate the safety profile of the maximum suitable dose. Optional treatment prolongations for 16 weeks (Amendment 2), 8 months (Amendment 3), 4 months (Amendment 4), and 12 months (Amendment 5).

Part 3- rapid dose escalation scheme from 6 mg to 720 mg of Talineuren followed by multiple doses of 720mg Talineuren for up to 8 months in 10 patients (Amendment 3).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature.
* Confirmed Parkinson's disease according to British brain bank criteria.
* Hoehn and Yahr Stage 0 - 2.5 on medication.
* Stable on PD treatment for a month at least.
* Absence of dementia confirmed by cognitive testing (MoCA >25).

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g., known hypersensitivity or allergy to class of drugs or the investigational product.
* Women who are pregnant or breast feeding, or planning to become pregnant during the course of the trial or in the 3 months following the trial.
* Lack of safe contraception in women with childbearing potential
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc) that is not under stable control.
* Subject has an atypical parkinsonian syndrome or secondary parkinsonism.
* Patients with comorbidity that may interfere with the course of the trial.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Occurence of adverse events (safety) | 8 to 134 weeks
  Number and kinds of adverse events (AEs)
Occurence of serious adverse events (safety) | 8 to 134 weeks
  Number and kinds of serious adverse events (SAEs)
Occurence of other safety-related signs (safety) | 8 to 134 weeks
  Number and kinds of other safety-related signs

SECONDARY OUTCOMES:
Levodopa challenge (LDC) test | 8 to 134 weeks
  Assessing the patients' condition via the LDC test (MDS-UPDRS-3 score)
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 8 to 134 weeks
  Assessing the patients' condition via the test
Epworth Sleepiness Scale (ESS) | 8 to 134 weeks
  Assessing the patients' condition via the test
Parkinson's Disease Questionnaire (PDQ-39) | 8 to 134 weeks
  Assessing the patients' condition via the test
Change in Parkinson's medication | 8 to 134 weeks
  Assessing the patients' condition via the change in their pre-existing Parkinson's medication
Starkstein Apathy Scale (SAS) | 8 to 134 weeks
  Assessing the patients' condition via the test
Montreal Cognitive Assessment (MoCA) | 8 to 134 weeks
  Assessing the patients' condition via the test
Beck's Depression Inventory (BDI) | 8 to 134 weeks
  Assessing the patients' condition via the test
Non-Motor Symptoms Questionnaire (NMSQuest) | 8 to 134 weeks
  Assessing the patients' condition via the test
Maximum Observed Drug Concentration (Cmax) in serum | 8 to 15 weeks
  Pharmacokinetics (PK) of total GM1 in serum over the first 96 h
Time of Maximum Drug Concentration (Tmax) in serum | 8 to 15 weeks
  Pharmacokinetics (PK) of total GM1 in serum over the first 96 h
Area Under the Curve to infinity (AUCinf.) in serum | 8 to 15 weeks
  Pharmacokinetics (PK) of total GM1 in serum over the first 96 h
half-life (t1/2) | 8 to 15 weeks
  Pharmacokinetics (PK) of total GM1 in serum over the first 96 h
Clearance (CL) | 8 to 15 weeks
  Pharmacokinetics (PK) of total GM1 in serum over the first 96 h
Volume of distribution (Vd) | 8 to 15 weeks
  Pharmacokinetics (PK) of total GM1 in serum over the first 96 h

CONTACTS AND LOCATIONS:
Locations (1):
- Neurologisches Institut Konolfingen, Konolfingen, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halbherr S, Lerch S, Bellwald S, Polakova P, Bannert B, Roumet M, Charles RP, Walter MA, Bernasconi C, Halbherr VL, Peitsch C, Baumgartner PC, Kaufmann C, Aires V, Mattle HP, Kaelin-Lang A, Hartmann A, Schuepbach M. Safety and tolerability of intravenous liposomal GM1 in patients with Parkinson disease: A single-center open-label clinical phase I trial (NEON trial). PLoS Med. 2025 May 13;22(5):e1004472. doi: 10.1371/journal.pmed.1004472. eCollection 2025 May. PMID 40359409
- [Derived] Roy R, Paul R, Bhattacharya P, Borah A. Combating Dopaminergic Neurodegeneration in Parkinson's Disease through Nanovesicle Technology. ACS Chem Neurosci. 2023 Aug 16;14(16):2830-2848. doi: 10.1021/acschemneuro.3c00070. Epub 2023 Aug 3. PMID 37534999